CLINICAL TRIAL: NCT05983601
Title: The Effect of Balance Training Combined With Motor Cortex Anodal Transcranial Direct Current Stimulation on Balance and Kinematic Parameters in Amateur Athletes
Brief Title: The Long-term Simultaneous Motor Cortex Stimulation and Balance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koc University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Marmara University (Other); İstinye University (Other)
Responsible Party: Principal Investigator, Ezgi Tuna Erdoğan, Ezgi Tuna Erdoğan, Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021.404.IRB.119; 321S329 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye)
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Coordination and Balance Disturbances
Keywords: Balance training; Transcranial Direct Current Stimulation; Neuromodulation; Non-invasive brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel controlled randomized double blind study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS+Balance training (Active Comparator): The current intensity will be 2mA and the duration of stimulation will be 20 minutes with direct current stimulation. In the beginning and end of the tDCS stimulation, there will be 30 second ascent and descent period.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS+Balance Training (Sham Comparator): In sham stimulation, the current will increase to 2 mA in the first thirty second, following by 30 second active stimulation, then it will be dropped to 0 mA. Brief electric current will be given in order to create a tingling sensation under electrodes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The anode electrode will be placed at the midline of the Cz according to international 10-20 EEG system, and the cathode electrode will be placed at the midline of forehead. In this way, both hemisphere of motor cortex can be stimulated which is used as protocol in various balance studies (Siedel-Marzi and Ragert, 2020b; Saruco et al., 2017). Participants will continue their training with tDCS (2mA) for 20 minutes. This application will continue three times a week for four weeks. In the end of the study, participants will be asked to guess which group they were in (active or sham).

SUMMARY:
Transcranial direct current stimulation (tDCS) is a simple, portable, and low-cost technology applied in neuroscience for therapeutic purposes and neurophysiological research of brain activity. Enhancing the impacts of training and improving performance in athletes through the use of tDCS is a significant aim for today.

The primary purpose of this study is to determine how non-professional active athletes' balance and movement measurements can be affected by the simultaneous application of a 4-week balance training and anodal tDCS of motor cortex(M1). This study hypothesizes that anodal stimulation of motor cortex will enhance performance in balance training among moderately active and healthy participants. The study outcomes will provide data for literatures on performance enhancement by demonstrating how effective skill development can be acquired in a short time among moderately active athletes. In addition, the study outcomes will provide convenient tDCS parameter for future neuromodulation studies interested in the treatment of balance disorders in patients and the elderly. Uniquely, in our study, the link between tDCS and movement parameters will be investigated. Additionally, a long-term balance training program in combination with tDCS of M1 in amateur has never been tested in amateur athletes.

The secondary purpose of the study is to obtain feedback from participants via pre- and post-tDCS and balance training, using continuous performance tests, estimated reaction time, and depression-anxiety scales to gather data on reaction time, anticipation, impulsivity, attention, and mood changes that directly affect athlete performance. In continuous performance test, a decrease in reaction times without an increase in the number of errors (misstep-commission) and the number of non-pressing (non-pressing-omission) will be considered as a successful outcome. While increasing balance performance and reducing the reaction time is anticipated as a positive outcome, simultaneously changes in mood, attention, and error rate is an unanticipated and undesired outcome. Although the selected stimulation area is not directly related to these functions, this study will additionally control for any potential changes that might have been missed in functions that are not the study's primary focus.

DETAILED DESCRIPTION:
Previous studies have demonstrated that the level of physical activity has an impact on response of tDCS application. While several studies found no tDCS effect on participants with both high and low levels of activity, it is expected to have greater impact on moderately active people. However, no study has yet investigated tDCS with moderately active athletes. Among studies investigating balance, only one study on healthy subjects has examined the correlation of tDCS implementation with kinematic parameters, and a correlation was found between increased balance performance and lower velocity parameter. By taking into account the effect of kinematic parameters on sports performance, this study intends to explore the effect of tDCS in greater detail by investigating both balance and movement analysis. This study will investigate the impact of combined anodal tDCS of motor cortex and 4-week balance-training program on static, dynamic balance and kinematic parameters in amateur athletes, and measure changes in reaction time and estimated reaction time. Previous studies showed that M1 anodal stimulation reduces reaction time, but estimated reaction time has never been examined. At the end of simultaneous tDCS-balance training, it is expected to reduce the reaction time without increasing the error rate and to achieve the expected reaction time, which is significant for improving athletes' performance.

Participants who met the requirements signed the informed consent form (BGOF) approved by the Ethics Committee and applied via the advertisements posted with permission from the university will be included in the study. Before the training and tDCS session, Beck Depression/ Anxiety Test and Dominant Foot Test will be applied to participants. Next, they will undergo a Continuous Performance Test (CPT) and an estimated reaction time test via a computer program and will last 5 minutes. CPT is a test performed to assess sustained attention and impulse control, where participants perform a task with a constant difficulty for several minutes. In addition, anthropometric measurements will be taken from the participants and these measures will be compared between sham and active groups to evaluate possible differences between two groups. After these tests, participants who are not suitable for the study will be eliminated, and remaining participants will be randomized into active or sham tDCS groups. Next, participants will attend a balance training session designed by a professional trainer to assess balance and movement parameters at the Koç University Movement Analysis Laboratory. The balance training program consists of a 5-minute warm-up and a 20-minute main section for the first and second weeks and a 5-minute warm-up and a 24-minute main section for the third and fourth weeks. The warm-up starts with a low-intensity cycling ergometer or low-intensity walking/running on a treadmill, followed by static/dynamic stretching exercises. During the 4-week balance training, the duration of a set is 30 seconds for the first two weeks and 45 seconds for the third and fourth weeks. Each exercise will be repeated twice on the right and left sides, totaling 4 repetitions. For some exercises, participants will perform them with their eyes open or closed, and on single or double legs. The tDCS device will be fixed on the participant's midline on their back and it will be constantly controlled during the training breaks and recharged if necessary. In case measurements cannot be taken due to a technical or scheduling issue, the same individuals will be recalled to the laboratory within the same week and they will be instructed not to engage in any extra training during that week.

At the end of 4-week combined balance training/ tDCS, participants will return to Movement Analysis Laboratory, and all tests performed at the beginning of study will be repeated. Individuals who miss two consecutive training sessions or a total of three training sessions in the 4-week program will be excluded from the study. To reduce the risk of this, participants will be provided with weekly schedules in advance. The next suitable participant identified through a pre-screening process will be included in place of those who are excluded from the study. Lastly, If the required number of participants cannot be reached during the initial interviews, the study announcement will be repeated and attempts will be made to recruit new participants. If sufficient participants cannot be provided from the Marmara University, amateur athletes who meet the research participant criteria will be sought outside of university.

ELIGIBILITY:
Inclusion Criteria:

* Scoring below 19 on the Beck Depression Inventory
* Scoring 15 or below on the Beck Anxiety Scale
* Having no neurological, psychiatric, orthopedic, or inner ear-related diseases
* Not being a professional athlete in a branch involving balance training (e.g., gymnastics)
* Not using medication affecting the central nervous system
* Having not consumed alcohol at least 24 hours prior to the tests
* Having no metal implants or hip/knee prosthesis
* Not being pregnant

Exclusion Criteria:

* Scoring 19 or higher on the Beck Depression Inventory
* Scoring higher than 15 on Beck Anxiety Scale
* Being a professional athlete
* Using mediation affecting the central nervous system
* Alcohol consumption less than 24 hours prior to the test
* Having metal implants or hip/knee prosthesis
* Being pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Dynamic Balance and Lower Extremity Functionality in Y-Balance Test Following 4-Week Simultaneous Balance Training and tDCS Treatment with 3 Sessions per week. | Baseline and Week 4
  The Y-balance test measures dynamic balance and the functionality of lower extremity. Participants perform reach tasks in 3 different directions with their legs and the maximum length reached is recorded before and after the tDCS treatment with simultaneous balance training. Scores are calculated by taking the sum of reach direction lengths, dividing by the length of upper extremity and multiplying by 100
  Change = (Week 4 Score - Baseline Score)
Changes from Baseline in BESS Scores Following a 4-Week Simultaneous Balance Training and tDCS Treatment with 3 Sessions per Week | Baseline and Week 4
  The Balance Error Scoring System is a standardized assessment tool that measures static balance and postural stability. In BESS, the number of errors or deviation from the normal stance is recorded, and changes in error are compared before and after tDCS treatment with simultaneous balance training.
  Change = (Week 4 Score - Baseline Score)
Changes from Baseline in Movement Parameters Recorded by Noraxon Myomotion 5 IMU Sensors During the Y-Balance test and BESS Movements Following a 4-Week Simultaneous Balance Training and tDCS Treatment with 3 Sessions per Week | Baseline and Week 4
  Noraxon Myomotion 5 IMU Sensors provide a detailed analysis of kinematics by quantifying motion and movement measures in various areas. These measures will be taken while participants perform Y-Balance and BESS movements. Change from baseline in Noraxon Myomotion 5 IMU Sensors parameters will allow for the interpretation of changes in precise movements performed in these tasks.
  Change = (Week 4 Score - Baseline Score)

SECONDARY OUTCOMES:
Changes from Baseline in Sustained Attention Measured by Continuous Performance Test Following a 4-Week Simultaneous Balance Training and tDCS Treatment with 3 Sessions per Week | Baseline and Week 4
  Continuous Performance Test is a well-known measurement to evaluate the sustained attention and response inhibition. Changes in omission and commission errors in CPT task will be compared before and after tDCS treatment with simultaneous balance training.
  Change = (Week 4 Score - Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Tuna Erdoğan, Principal Investigator — Koç University
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No